CLINICAL TRIAL: NCT03853980
Title: The INFORM Study: A Multi-Center Study to Evaluate the Safety and Efficacy of Rotational Fractional Resection on Submental Contouring With an Optimized Post-Procedure Treatment Plan
Brief Title: The INFORM Study: Rotational Fractional Resection for Submental Contouring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Recros Medica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-0006
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Skin Laxity
Keywords: submental; laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Rotational fractional resection (RFR) (Experimental): Single treatment of skin resection (removal of loose skin)
  Interventions: Device: Focal Contouring System

INTERVENTIONS:
Device: Focal Contouring System — Single treatment of skin resection (removal of loose skin)

SUMMARY:
Efficacy and safety of Rotational Fractional Resection (skin resection) in patients with moderate to severe submental skin laxity.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm (non-randomized), interventional cohort, non-significant risk (NSR) study designed to investigate the efficacy and safety of Rotational Fractional Resection (skin resection) in patients with moderate to severe submental skin laxity. The total duration of study participation for each subject is approximately up to 4 months for each subject from the screening visit to the exit visit. The follow-up period will be approximately 3 months after the procedure. Eligible subjects will complete a total of 11 study visits: screening, procedure, and follow-up visits at 1, 2-4, 7, 14, 21, 30, 45, 60, and 90 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* At least 30 years old
* Moderate to severe submental laxity
* Agree to maintain weight (±5%) for the duration of the study

Exclusion Criteria:

* Greater than mild submental fat
* Previous intervention to treat submental fat or skin laxity
* Use of aspirin, ibuprofen, naproxen, or Vitamin E within 14 days of the procedure
* Severe acne, cystic acne or acne scars on neck
* Trauma of chin or neck area
* Skin infection or rash on neck
* Psoriasis, hyperpigmentation, eczema, rosacea or vitiligo
* History of scarring
* Body mass index (BMI) >30
* Clinically significant bleeding disorder
* Anemia, kidney disease, or liver disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Improved Skin Laxity | Pre-treatment and 90 days after treatment
  Comparison of the submentum before and after procedure using the Submental Skin Laxity scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe)
Subject Satisfaction: Subject Satisfaction Questionnaire | Pre-treatment and 90 days after treatment
  Comparison of Subject satisfaction of the procedure as assessed using the Subject Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robin McIntosh, Study Director — Recros Medica
Locations (14):
- United States (14):
  - Aesthetx, Campbell, California
  - Clinical Testing of Beverly Hills, Encino, California
  - Westside Aesthetics, Los Angeles, California
  - ATS Clinical Research, Santa Monica, California
  - Moradi MD, Vista, California
  - AboutSkin Research, Greenwood Village, Colorado
  - Washington Institute of Dermatologic Laser Surgery, Washington D.C., District of Columbia
  - DeNova Research, Chicago, Illinois
  - Juva Skin and Laser Center, New York, New York
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Brian Biesman, MD, Nashville, Tennessee
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Sundaram Dermatology, Cosmetic & Laser Surgery Center, Fairfax, Virginia
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No